CLINICAL TRIAL: NCT01155440
Title: Restoration of Bowel Function After Laparoscopic Colorectal Surgery: Effect of Intravenous Lidocaine
Brief Title: Bowel Function After Laparoscopic Colon Surgery: Effect of IV Lidocaine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gabriele Baldini, Assistant Professor, Dr, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GEN-06-023(1)
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Colon Cancer; Inflammatory Bowel Diseases; Diverticulitis
Keywords: 60 patients scheduled to have a colorectal surgery; recruit at Montreal General Hospital
MeSH Terms: conditions — Colonic Neoplasms; Inflammatory Bowel Diseases; Diverticulitis | interventions — Lidocaine; Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LIDOCAINE group (Experimental): Beside general anesthesia, patients will receive intravenous lidocaine bolus 1.5 mg/kg just prior induction and an infusion of lidocaine 2mg/kg/h will be started and maintained during the whole surgical procedure. Entering the recovery room, this infusion will be decreased at the rate of 1mg/kg/hour for the 48 first hours
  Interventions: Drug: Lidocaine
- Epidural group (Active Comparator): Beside general anesthesia, patient will receive epidural freezing medication for 48 hours.
  Interventions: Procedure: Thoracic epidural block

INTERVENTIONS:
Drug: Lidocaine — 1% Lidocaine 1mg/kg/hr IV drip x 48hr
  Other Names: Xylocaine
  Arms: LIDOCAINE group
Procedure: Thoracic epidural block — 0.1% Epidural bupivacaine + Morphine 0.02 mg/ml drip via epidural x48 hr
  Other Names: Thoracic Epidural analgesia
  Arms: Epidural group

SUMMARY:
Patients receiving perioperative intravenous lidocaine, post operative restoration of bowel movement will be faster and decrease pain intensity, opioid consumption and side effects, length of hospital stay; probably as a result of a significant opioid sparing and attenuated inflammatory response.

DETAILED DESCRIPTION:
The aim of this study is to assess whether perioperative intravenous lidocaine has an impact on the early postoperative physical activity recovery of patients scheduled for laparoscopic colorectal resection.

The study focuses on patients with colorectal disease, which receive the laparoscopic (assisted) surgical approach.

It is hypothesized that in those patients receiving perioperative and post-operative intravenous lidocaine, bowel function recovery will be faster, probably as a result of a significant opioid sparing, less pain and attenuated inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo laparoscopic colorectal resection

Exclusion Criteria:

* patients who have trouble to understand, read or communicate either in French or in English
* dementia
* patients suffering from severe physical disability (arthritis, neuromuscular dysfunction, stroke, paraplegia) or inability to walk or conduct daily activity
* patients suffering from severe cardiac or respiratory disease (status ASA IV
* patients suffering from metastatic carcinoma
* patients who have a history of chemoradiation within the six months preceding surgery
* allergy to lidocaine
* morbid obesity
* patients with chronic opioid use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Restoration of bowel function | 72 hours after an operation

SECONDARY OUTCOMES:
Pain intensity | within 72 hours after an operation
  Visual analog score pain (from 0-10) at rest, on walking and coughing at 24, 48 and 72 hours after an operation are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, Fellow, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- MUHC, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Wongyingsinn M, Baldini G, Charlebois P, Liberman S, Stein B, Carli F. Intravenous lidocaine versus thoracic epidural analgesia: a randomized controlled trial in patients undergoing laparoscopic colorectal surgery using an enhanced recovery program. Reg Anesth Pain Med. 2011 May-Jun;36(3):241-8. doi: 10.1097/AAP.0b013e31820d4362. PMID 21519309